CLINICAL TRIAL: NCT01870947
Title: REWARD (Revving-Up Exercise for Sustained Weight Loss by Altering Neurological Reward and Drive): A Randomized Trial of Assisted Exercise in Obese Endometrial Cancer Patients
Brief Title: Assisted Exercise in Obese Endometrial Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5811
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Stage I Endometrial Adenocarcinoma; Uterine Cancer; Obesity
Keywords: Stage I endometrial adenocarcinoma; Obesity; Exercise and Physical Fitness; Diet; Cancer
MeSH Terms: conditions — Uterine Neoplasms; Obesity; Motor Activity; Neoplasms | interventions — Surveys and Questionnaires; Neuroimaging; Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Assisted-Rate' Exercise Intervention (Experimental): Subjects in the assisted exercise group will cycle on the same stationary exercise bike; however, a motor will provide assistance to the patient in order to maintain a pedaling rate 35% greater than their voluntary rate. Subjects in the exercise groups will complete 45 minute to 1-hour sessions, three times per week for eight weeks.
  Interventions: Behavioral: Exercise on stationary recumbent exercise cycle; Behavioral: Health Education; Behavioral: Questionnaires; Procedure: Neuroimaging; Procedure: Genetic and Biomarkers
- 'Voluntary-Rate' Exercise Intervention (Experimental): Subjects in the voluntary group will exercise on a stationary recumbent exercise cycle and pedal at their preferred rate. Subjects in the exercise groups will complete 45 minute to 1-hour sessions, three times per week for eight weeks.
  Interventions: Behavioral: Exercise on stationary recumbent exercise cycle; Behavioral: Health Education; Behavioral: Questionnaires; Procedure: Neuroimaging; Procedure: Genetic and Biomarkers

INTERVENTIONS:
Behavioral: Exercise on stationary recumbent exercise cycle
Behavioral: Health Education — Informational brochure ("Better Health and You," Weight Control Information Network, June, 2004)
Behavioral: Questionnaires
  Other Names: Exercise Motivations Inventory (EMI-2); Intrinsic Motivational Inventory (IMI); Three-Factor Eating Questionnaire (TFEQ); Functional Assessment of Cancer Therapy - General (FACT-G); FACT-En; Short-form Medical Outcomes (SF-36); Beck Depression Inventory (BDI); Godin Leisure-Time Exercise (LSI)
Procedure: Neuroimaging — Imaging data will be acquired on a Siemens 3.0T Wide-Bore Verio MRI scanner.
  Other Names: MRI
Procedure: Genetic and Biomarkers — Patients will be asked to fast for approximately 12 hours and will have approximately 2 Tbs. of blood drawn at baseline and the end of treatment (EOT).
  Other Names: DNA Testing; Biomarker Testing

SUMMARY:
This is an assisted exercise trial involving exercise on a stationary bike, brain imaging and DNA(genetics)sampling. The purpose of this study is to find out if performing a progressive, supervised assisted exercise program on a stationary bike improves quality of life, increases motivation to continue to exercise, improves dietary behavior and leads to sustained weight loss in women who have had early-stage endometrial cancer. Questionnaires will be used to assess exercise motivation and dietary behavior. Brain's responses to different visual images will also be assessed.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate changes in body weight, fitness, bi-manual dexterity, exercise motivation and self-reported eating behavior (via questionnaires) before and after a 16-week exercise intervention (EOT) and 12 and 24 weeks post-EOT, in obese EC patients who will be randomized to perform 'assisted' or voluntary exercise.

Secondary Objectives:

Objective 1: To objectively examine food behavior as determined by neuronal response to high- versus low-calorie visual stimuli under fasted (hunger) and fed (satiated) states and stop/go signaling (SST) in fed states in brain regions of interest (reward and motivation circuitry) using blood oxygenation level dependent (BOLD) functional MRI before and after a 16-week exercise intervention (EOT) and 12 and 24 weeks post-intervention in obese EC patients performing 'assisted' and voluntary exercise.

Objective 2: To examine the modification of the neuronal response to high vs. low calorie food images in regions of interest by polymorphisms in key genes (e.g., dopamine receptor and dopamine transporter) and serum biomarkers (e.g., leptin, BDNF) involved in regulating homeostatic and non-homeostatic energy systems.

Patients will be randomized to receive either the assisted exercise (n=60) or voluntary exercise (n=60) group. Subjects in the voluntary group will exercise on a stationary recumbent exercise cycle and pedal at their preferred rate. Subjects in the assisted exercise group will cycle on the same stationary exercise bike; however, a motor will provide assistance to the patient in order to maintain a pedaling rate 35% greater than their voluntary rate. Subjects in the exercise groups will complete 45 minute to 1-hour sessions, three times per week for eight weeks. The control group will be asked to complete all exercise, body composition and fMRI testing similar to the exercise groups.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage I endometrial adenocarcinoma (EC), grade 1 or 2, with no adjuvant chemotherapy. Patients will be eligible to enroll as soon as 3 months after completion of treatment but no later than 4 years after completion of treatment.
* BMI ≥ 30.0 (obese)
* Approved to be contacted by the patient's treating gynecologic oncologist
* Meets screening criteria including successful completion of a cardiopulmonary stress test
* Receives medical clearance from the patient's primary care physician (PCP) or gynecologic oncologist to exercise in this study

Exclusion Criteria:

* Individuals unable to read and provide informed consent.
* Women currently participating in a structured weight loss or exercise program in the past 6 months or any woman who has previously had bariatric surgery or is planning to undergo bariatric surgery in the next 12 months
* Participants who do not consent to be in the study or who will be unavailable for follow-up assessments,
* Pre-existing medical conditions that would be a barrier for participation in supervised exercise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-09-07 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Weight change from pre- to post-intervention | 24 weeks after exercise intervention (EOT)

SECONDARY OUTCOMES:
Change in Body Composition from baseline | at 4 weeks after exercise intervention(EOT)
  Body fat, lean mass and bone mass will be measured with a Lunar iDXA™ (GE Healthcare, Madison, WI. BMI will be computed (weight in kg divided by square of height in meters) and categorized as: < 18.5 (underweight), 18.5 to 24.9 (normal weight), 25.0 to 29.9 (overweight)
Change in Motivation to Exercise from baseline | 24 weeks after exercise intervention (EOT)
  Evaluate motivation to exercise using the Exercise Motivations Inventory (EMI-2) 122 and the Intrinsic Motivational Inventory (IMI) modified for exercise. Past physical activity habits will be assessed with the Godin Leisure-Time Exercise (LSI) questionnaire.
Change in Eating Behavior from baseline | 24 weeks after exercise intervention (EOT)
  Eating behavior will be assessed using the Three-Factor Eating Questionnaire (TFEQ). The TFEQ includes 51 items and addresses three dimensions of human eating behavior; restraint, disinhibition, and perceived hunger.
Change in Quality of Life (QoL)from baseline | 24 weeks after exercise intervention (EOT)
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item core questionnaire evaluating various domains of QoL including, physical, functional, family-social, and emotional well-being. The FACT-En is a 16-item subscale specific for endometrial cancer (EC) and assesses hormone withdrawal, pelvic symptoms, and possible adjuvant therapy side effects. Short-form Medical Outcomes (SF-36) consists of 36 questions scored on a Likert scale, producing overall physical and mental component summary measures.
Change in Depression from baseline | 24 weeks after exercise intervention (EOT)
  The Beck Depression Inventory (BDI) is a 21-item, Likert-scaled instrument of depressive symptoms that is well-validated and frequently used in lifestyle research studies. Each item is rated on a 4- point scale ranging from 0 to 3 (higher scores are associated with greater symptoms).
Exercise Session Adherence | 24 weeks after exercise intervention (EOT)
  Barriers to adhering to the exercise protocol will be assessed prospectively using an elicitation procedure similar to that suggested in the theory of planned behavior, whereby an open-ended question is asked to solicit the barrier without any preconceived notion of what the barrier might be. Specifically, participants in the exercise groups will be asked to book their weekly supervised exercise sessions with the Exercise Specialist/Physiologist. Participants cancelling an exercise session or requesting to be removed from the study will be asked why they are no longer interested in completed the program.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Nock, PhD, Principal Investigator — Cleveland Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Cleveland Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Derived] Nock NL, Dimitropoulos A, Zanotti KM, Waggoner S, Nagel C, Golubic M, Michener CM, Kirwan JP, Alberts J. Sleep, quality of life, and depression in endometrial cancer survivors with obesity seeking weight loss. Support Care Cancer. 2020 May;28(5):2311-2319. doi: 10.1007/s00520-019-05051-1. Epub 2019 Sep 2. PMID 31478164